CLINICAL TRIAL: NCT01838915
Title: Gut Microbiota, Bacterial Translocation, Immune Activation and Endothelial Dysfunction in HIV Infection
Brief Title: Randomized Placebo-controlled Pilot Trial of Prebiotics+Glutamine in HIV Infection
Acronym: MicroVIH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Sergio Serrano-Villar, Post-Doctoral Researcher, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/284
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: HIV
Keywords: HIV; immunoactivation; bacterial translocation; prebiotics; glutamine; microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Supplement: Prebiotics+Glutamine (Experimental)
  Interventions: Dietary Supplement: Prebiotics+Glutamine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotics+Glutamine — Prebiotics are nondigestible food ingredients, generally oligosaccharides, that modify intestinal microbiota balance by stimulating the growth of beneficial bacteria.
  Glutamine is a non-essential amino acid that can be metabolized by epithelial cells, enhancing barrier function.
  Arms: Dietary Supplement: Prebiotics+Glutamine
Dietary Supplement: Placebo — Maltodextrin, 20 g.
  Arms: Placebo

SUMMARY:
A rapid and almost complete loss of CD4+ T cells from the gut associated lymphoid tissue (GALT) occurs early in HIV infection, with a permanent damage in the intestinal barrier, changes in gut microbiota, increased bacterial translocation and persistent immune activation, changes that are not restored after the initiation of antiretroviral therapy. The investigators hypothesize than an intervention targetting the enterocyte barrier and the gut microbiota might modify the gastrointestinal tract towards a bifidogenic microbiota and improve markers of bacterial translocation, inflammation, immune activation and endothelial dysfunction.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled clinical trial to evaluate the safety and effectiveness to modify gut microbiota, bacterial translocation, immune activation and markers of endothelial dysfunction of a dietary supplement (prebiotics + glutamine) during a period of six weeks. The study will enroll four cohorts: 1) HIV-infected, treatment naive individuals; 2) HIV-infected subjects, currently on ART, with >350 CD4+ T-cells/uL; 3) HIV-infected subjects, currently on ART, with <350 CD4+ T-cells/uL; 4) HIV negative healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* After receiving information on the design and objectives of the study, the possible risks involved, and the fact that they can refuse to collaborate at any time, patients will give their informed consent to participate in the study and agree to provide material for the cellular and molecular studies.
* Aged over 18 years.
* Group 1: HIV+, Not receiving ART and no previous exposure to ART, at least 2 years since HIV diagnosis.
* Group 2: HIV+, currently receiving ART for more than 2 years, HIV-1 RNA levels less than 40 copies/ml and more than 350 CD4+ T-cells/uL.
* Group 3: HIV+, currently receiving ART for more than 2 years, HIV-1 RNA levels less than 40 copies/ml and less than 350 CD4+ T-cells/uL.
* Group 4: HIV-, healthy controls.

Exclusion Criteria:

* Major cardiovascular risk factors.
* Concomitant acute diseases.
* Gastrointestinal disorders.
* Pregnancy.
* Antibiotic exposure in the previous month.
* Regular use of foods or supplements containing prebiotics or probiotics within the 2 weeks prior to initiation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Safety | 6 weeks
  Adverse events monitoring during the intervention
Changes in markers of bacterial translocation | 6 weeks
  Soluble CD14 and increasing permeability binding protein.
Changes in markers of immunoactivation | 6 weeks
  Changes in percentages of CD4+ and CD8+ T-cells expressing CD25, HLADR, CD38.
Changes in inflammatory markers | 6 weeks
  Changes in interleukine-6 and high-sensitivity C Reactive Protein
Changes in markers of endothelial dysfunction | 6 weeks
  Changes in asymmetric dimethylarginine and flow-mediated dilation
Changes in gut microbiota composition | 6 weeks
  Changes in gut microbiota as determined by 454 pyrosequencing.

SECONDARY OUTCOMES:
Changes in gut microbiota | 6 weeks
  Changes in gut microbiota by 454 pyrosequencing of fecal samples.
Disease progression in HIV-infected patients. | 6 weeks
  Levels of CD4+ T-cell and HIV-1 RNA copies/mL
Thymic function | 6 weeks
Gene expression in peripheral blood monocytic cells. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal and Hospital Clínico San Carlos, Madrid, Spain